CLINICAL TRIAL: NCT01777022
Title: Promoting Awareness Fetal Movements and Focussing Interventions Reduce Fetal Mortality Stillbirth, a Stepped Wedge Cluster Randomised Trial.
Brief Title: Promoting Awareness Fetal Movements to Reduce Fetal Mortality Stillbirth, a Stepped Wedge Cluster Randomised Trial.
Acronym: AFFIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: AFFIRM
Record Dates: First submitted 2013-01-15; First posted 2013-01-28 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Decreased Fetal Movements Affecting Care of Mother; Pregnancy; Stillbirth
Keywords: Education, Stillbirth, Prevention, Management
MeSH Terms: conditions — Stillbirth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Current treatment (No Intervention): Current education and management protocols will be followed
- A package of interventions (Other): A package of interventions consisting of strategies for increasing pregnant women's awareness of the need to report early when they perceive a reduction in fetal movements, followed with a management plan for identification and delivery of the "at risk" fetus in such women, will reduce rates of stillbirth
  Interventions: Other: A package of interventions

INTERVENTIONS:
Other: A package of interventions — A package of interventions consisting of strategies for increasing pregnant women's awareness of the need to report early when they perceive a reduction in fetal movements, followed with a management plan for identification and delivery of the "at risk" fetus in such women, will reduce rates of stillbirth
  Arms: A package of interventions

SUMMARY:
Rates of stillbirth in Scotland are among the highest in resource rich countries. The majority of stillbirths occur in normally formed infants, with (retrospective) evidence of placental insufficiency being the commonest clinical finding. Maternal perception of decreased fetal movements appears to be an early biomarker both of placental insufficiency and subsequent stillbirth.

The study proposed here will test the hypothesis that rates of stillbirth will be reduced by introduction of a package of care consisting of strategies for increasing pregnant women's awareness of the need for prompt reporting of decreased fetal movements, followed by a management plan for identification of placental insufficiency with timely delivery in confirmed cases. The odds of stillbirth fell by 30% after the introduction of a similar package of care in Norway but the efficacy of this intervention (and possible adverse effects and implications for service delivery) have not been tested in a randomized trial.

The investigators plan a stepped wedge cluster design trial, in which hospitals in Scotland and Ireland will be randomized to the timing of introduction of the care package. Outcomes (including the primary outcome of stillbirth) will be derived from Scotland and Ireland's detailed routinely collected maternity data, allowing the investigators to robustly test the hypothesis. A nested qualitative study will examine the acceptability of the intervention to patients and health care providers and identify process issues (barriers to implementation).

ELIGIBILITY:
Inclusion Criteria:

* The study will include all women delivering at one of the maternity units involved in for the duration of the study.

Exclusion Criteria:

* Women delivering in the "washout" period in each unit.

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 430830 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Rates of stillbirth | 36 months

SECONDARY OUTCOMES:
Rates of caesarean section | 36 months
Rates of induction of labour | 36 Months
Rates of admission to the neonatal intensive care unit | 36 Months
Proportion of women with fetal growth restriction | 36 Months

OTHER OUTCOMES:
Acceptability of package of care to pregnant women and their health care providers | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Norman, MD, Study Chair — University of Edinburgh
Locations (29):
- Ireland (2):
  - National Maternity Hospital, Dublin
  - Rotunda Hospital, Dublin
- United Kingdom (27):
  - Stepping Hill Hospital, Stockport, Cheshire
  - Royal Gwent Hospital, Newport, Gwent
  - Saint Mary's hospital, Manchester, Lancashire
  - NHS Lothian, Edinburgh, Lothian
  - Birmingham Women's Hospital, Birmingham, West Midlands
  - St. Richards Hospital, Chichester, West Sussex
  - Worthing Hospital, Worthing, West Sussex
  - Leeds Teaching Hospital NHS Trust, Leeds, Yorkshire
  - NHS Grampian, Aberdeen
  - Neville Hall hospital, Abergavenny
  - Betsi Cadwaladr University Heath board (Ysbyty Gwynnedd Hospital), Bangor
  - Royal Jubilee Hospital, Belfast
  - Blackpool Victoria Hospital, Blackpool
  - NHS Dumfries and Galloway, Dumfries
  - NHS Tayside, Dundee
  - NHS Greater Glasgow, Glasgow
  - NHS Highland, Inverness
  - NHS Ayrshire and Arran, Kilmarnock
  - NHS Fife, Kirkcaldy
  - NHS Forth Valley, Larbert
  - St Georges Hospital, London
  - NHS Borders, Melrose
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Betsi Cadwaladr University Heath board (Glan Clwyd), Rhyl
  - Royal Albert Edward Infirmary, Wigan, Wigan
  - NHS Lanarkshire, Wishaw
  - Betsi Cadwaladr University Heath board (Wrexham Maelor), Wrexham

REFERENCES:
- [Derived] Camacho EM, Whyte S, Stock SJ, Weir CJ, Norman JE, Heazell AEP. Awareness of fetal movements and care package to reduce fetal mortality (AFFIRM): a trial-based and model-based cost-effectiveness analysis from a stepped wedge, cluster-randomised trial. BMC Pregnancy Childbirth. 2022 Mar 22;22(1):235. doi: 10.1186/s12884-022-04563-9. PMID 35317772
- [Derived] Norman JE, Heazell AEP, Rodriguez A, Weir CJ, Stock SJE, Calderwood CJ, Cunningham Burley S, Froen JF, Geary M, Breathnach F, Hunter A, McAuliffe FM, Higgins MF, Murdoch E, Ross-Davie M, Scott J, Whyte S; AFFIRM investigators. Awareness of fetal movements and care package to reduce fetal mortality (AFFIRM): a stepped wedge, cluster-randomised trial. Lancet. 2018 Nov 3;392(10158):1629-1638. doi: 10.1016/S0140-6736(18)31543-5. Epub 2018 Sep 27. PMID 30269876
- [Derived] Heazell AEP, Weir CJ, Stock SJE, Calderwood CJ, Burley SC, Froen JF, Geary M, Hunter A, McAuliffe FM, Murdoch E, Rodriguez A, Ross-Davie M, Scott J, Whyte S, Norman JE. Can promoting awareness of fetal movements and focusing interventions reduce fetal mortality? A stepped-wedge cluster randomised trial (AFFIRM). BMJ Open. 2017 Aug 11;7(8):e014813. doi: 10.1136/bmjopen-2016-014813. PMID 28801392

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT01777022/SAP_000.pdf
  • Study Protocol (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT01777022/Prot_001.pdf